CLINICAL TRIAL: NCT01099488
Title: A Study in Healthy Adults Having Received a Single Vaccine Administration to Support the Development of Immunological Assays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113737
Record Dates: First submitted 2010-03-26; First posted 2010-04-07 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Immunologic Tests
Keywords: Immunological assays

ARMS (1):
- All subjects (Other): Healthy male or female adults between, and including, 18 and 50 years of age at the time of study start, having received a GSK2231392A vaccine, were enrolled for blood withdrawal to support the development of CD8+ T cell immunological detection assays.
  Interventions: Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Blood withdrawal — Healthy male or female adults between, and including, 18 and 50 years of age at the time of study start, having received GSK2231392A vaccine, were enrolled for blood withdrawal, at each study visit: Day 0, Day 14 and Day 180, to support the development of CD8+ T cell immunological detection assays.

SUMMARY:
The purpose of this study is to develop immunological assays on blood samples.

DETAILED DESCRIPTION:
This is a clinical study in which there is no vaccine administered. It is designed for research purposes such as developing immunological assays.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol (e.g. return for follow-up visits).
* A male or female between, and including, 18 and 50 years of age at study start.
* A subject having received a Yellow Fever (YF) vaccine on the day of study entry.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination performed on the day of YF vaccination.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to study start, and
  * has agreed to continue adequate contraception during the entire study period.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding study start, or planned use during the study period.
* Concurrently participating in another clinical study, within 3 months preceding study start and at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Clinically significant anaemia or any known condition as per medical history that would preclude the drawing of blood as described in the protocol.
* Known previous infection with YF virus.
* Previous vaccination against YF more than approximately 5 hours before the blood sampling at Visit 1.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the study start or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs (including chloroquine) within six months prior to the study start. For corticosteroids, this will mean prednisone ≥ 10mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Receipt of live attenuated vaccines other than the YF vaccine during the period beginning 30 days preceding the blood sampling at Visit 1 or planned use during the study up to the blood sampling at Visit 2.
* Receipt of inactivated influenza vaccines (seasonal or pandemic) during the period beginning 21 days preceding the blood sampling at Visit 1 or planned use during the study up to the blood sampling at Visit 2.
* History of malignancy (unless there has been surgical excision followed by a sufficient observation period, of at least 5 years, to give a reasonable assurance of sustained cure and which, in the estimate of the investigator, is not likely to recur during the study period).
* Any confirmed or suspected immunosuppressive or immunodeficient condition (including HIV, hepatitis B and hepatitis C), based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination and medical history.
* Acute disease and/or fever at the time of enrolment.
* Known pregnant or lactating female, as per medical records.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Any condition that may preclude the compliance to the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2010-04-01; Primary Completion 2010-12-07 (Actual); Study Completion 2010-12-07 (Actual)

PRIMARY OUTCOMES:
Frequency of CD8+ T-cells at protocol-defined time points. | At Day 0, Day 14 and Day 180.

SECONDARY OUTCOMES:
Frequency of CD4+ T-cells response at protocol-defined time points. | At Day 0, Day 14 and Day 180.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Belgium (2):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Mons